CLINICAL TRIAL: NCT00876850
Title: A Randomized, Evaluator-Blinded, Phase 3 Study to Compare the Safety and Efficacy of PTK 0796 With Linezolid in the Treatment of Adults With Complicated Skin and Skin Structure Infection
Brief Title: Phase 3 Study - Safety and Efficacy of PTK 0796 in Patients With Complicated Skin and Skin Structure Infection (CSSSI)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTK 0796-CSSI-0805
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Skin Structures and Soft Tissue Infections
Keywords: cSSI; Abscess; Would; Cellulitis; Complicated Skin and Skin Structure Infections (cSSSI)
MeSH Terms: conditions — Soft Tissue Infections; Abscess; Cellulitis | interventions — 7-dimethylamino-9-(2,2-dimethylpropyl)aminomethylcycline; Linezolid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTK 0796 (Experimental): PTK 0796 100mg for injection; PTK 0796 tablet 150mg
  Interventions: Drug: PTK 0796
- Linezolid (Active Comparator): For gram positive treatment: Linezolid 600 mg tablets and pre-mixed 600mg IV infusion solution; For gram negative treatment: Moxifloxacin 400 mg tablets and pre-mixed 400mg IV infusion solution
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: PTK 0796 — PTK 0796 100mg for injection; PTK 0796 tablet 150mg
  Arms: PTK 0796
Drug: Linezolid — For gram positive treatment: Linezolid 600 mg tablets and pre-mixed 600mg IV infusion solution; For gram negative treatment: Moxifloxacin 400mg tablets and pre-mixed 400mg IV infusion solution
  Other Names: Zyvox™; Avelox™
  Arms: Linezolid

SUMMARY:
A Phase III trial to demonstrate the safety and efficacy of PTK 0796 in the treatment of complicated skin and skin structure infections (cSSSI).

DETAILED DESCRIPTION:
The pharmacologic profile of PTK 0796 in humans suggests that it has the potential to be used safely and effectively for this indication. Data from in vitro and animal studies support this hypothesis.

In PTK 0796-CSSI-0805 the safety and efficacy of PTK 0796 in the treatment of cSSSI will be compared to an antibiotic approved for this indication by the FDA. Initial treatment will be administered intravenously with the option for subsequent oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has and acute complicated skin and skin structure infection with findings of systemic inflammatory response
* Patients, ages 18 years or older
* Is expected to require greater than or equal to 4 days antibiotic therapy
* Female patients must not be pregnant at the time of enrollment and must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Has received an investigational drug within the past 1 month
* Has been previously enrolled in this protocol
* Has received >48hr of potentially effective systemic antibiotic immediately prior to study drug
* Is nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Clinical success at follow-up | 4 weeks after enrollment

SECONDARY OUTCOMES:
To evaluate safety of dosing regimens | 4 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Arbeit, MD, Study Director — Paratek Pharmaceuticals Inc